CLINICAL TRIAL: NCT04474496
Title: Impact of COVID-19 on Marshallese Communities in the U.S.
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 261131
Record Dates: First submitted 2020-07-10; First posted 2020-07-16 (Actual); Results first posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
Keywords: Marshallese; Pacific Islanders; Type 2 Diabetes; COVID-19
MeSH Terms: conditions — COVID-19; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Marshallese adults in the U.S.: Marshallese persons 18 years of age or older currently residing in the United States
  Interventions: Other: Assessing the impact of COVID-19

INTERVENTIONS:
Other: Assessing the impact of COVID-19 — Surveying Marshallese adults in the U.S. to determine the impact of COVID-19

SUMMARY:
Marshallese adults in the U.S. will complete an online or telephone survey. This survey will collect data describing the impact of COVID-19 on Marshallese communities. Data collected will help describe: 1) risk exposure, 2) knowledge of preventive recommendations, 3) barriers and facilitators to implementing preventative recommendations, 4) barriers and facilitators to COVID-19 testing when appropriate, and 5) self-care behaviors during COVID-19. Participant inclusion criteria: 1) Self-reported Marshallese; 2) 18 years of age or older; 3) Live in the Continental U.S. or Hawaii.

DETAILED DESCRIPTION:
Background and Rationale

While there is much we do not know about the differential effects of COVID-19, early data shows that minority communities are disproportionally effected by the virus. There are many factors that may increase the likelihood of contracting COVID-19 including: 1) community spread because of lack of access to testing in low-income communities, 2) work environments that may increase exposure, 3) more densely populated housing that reduces the ability to social distance, 4) limited understanding of preventive measures due to literacy and language barriers, 5) constrained financial resources to stay home and not work, and/or 6) lack of trust in the health care system. The Marshallese are a Pacific Islander population experiencing significant health disparities with some of the highest documented rates of type 2 diabetes mellitus (T2DM) of any population in the world. Estimated T2DM rates among Marshallese in the U.S. range from 25%-50%, much higher than the general U.S. population. People with T2DM are more likely to experience severe symptoms and complications when infected with COVID-19; however, those that manage their T2DM well are less likely to become extremely ill from the virus. In order to reduce the disparities caused by COVID-19 and ultimately compare the effectiveness of prevention interventions among the low-income minority communities most effected by COVID-19, it is critical to understand minority populations': 1) risk exposure, 2) knowledge of preventive recommendations, 3) barriers and facilitators to implementing preventative recommendations, 4) barriers and facilitators to COVID-19 testing when appropriate, and self-care behaviors during COVID-19.

Specific Aims

Aim 1: Document COVID-19 risk exposure for Marshallese community members.

Aim 2: Document Marshallese community members' knowledge of preventive recommendations.

Aim 3: Document barriers and facilitators to implementing preventative recommendations.

Aim 4: Document Marshallese community members' barriers and facilitators to COVID-19 testing when appropriate.

Aim 5: Document self-care behaviors during COVID-19.

Aim 6: Explore COVID-19 pandemic related barriers and facilitators to T2DM self-management among Marshallese adults with T2DM.

Aim 7: Assess the effect of the COVID-19 pandemic on T2DM self-management activities among Marshallese adults with T2DM.

Study Design and Procedures

Participants will complete an online or telephone survey. Up to 100 participants will also be invited to complete an in-depth qualitative interview in addition to the survey (these results are not presented here). Community-based recruitment for the online survey will be conducted by posting an informational flyer on social media. The flyer will contain a link to the study information sheet and survey documents. Study team members will also reach out to study participants via phone or electronic mediums (e.g. email, text, or messenger). Study staff will send potential participants a link to an electronic survey using REDcap. The REDcap system will include electronic documentation of consent prior to completing the survey. Access to study data will be limited to only those personnel who need it to complete relevant job duties. All data, regardless of whether it is identifiable or not, will be stored in a locked file cabinet in a locked room, or on a secure University of Arkansas for Medical Sciences (UAMS) server that requires two-factor authentication.Each participant who completes the survey will receive a $20 Walmart gift card as remuneration.

Measures/outcomes

Our survey will be based on CDC risk assessments and utilize the NIH funded COVID-19 items that are part of the PhenX Toolkit, as well as other standardized survey items/scales. Those participants with T2DM will be asked to complete questions pertaining to T2DM self-management during COVID-19.

Data Analysis

Given the descriptive nature of the study aims, the analytic strategy will focus on presenting results of item-level descriptive analyses, with an emphasis on frequencies and proportions. There will be no attempt to impute missing responses for any items. For each analysis, the number of included responses will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Marshallese
* 18 years of age or older
* Live in the Continental U.S. or Hawaii

Exclusion Criteria:

- Does not meet inclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Self-reported Marshallese persons 18 years of age or older who live in the continental United States or Hawaii.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pearl A McElfish, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences Northwest, Fayetteville, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was open from July 27, 2020 to November 30, 2020. The study was advertised by posting informational flyers on social media. Flyers contained a link to the study information sheet and survey.
Period: Overall Study
Arm/Group | Marshallese Adults in the U.S.
Started | 120
Completed | 120 (120 individuals were deemed eligible based on inclusion criteria, completed at least 10 survey items, and were included in the final analytical sample)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 120 eligible individuals completed at least 10 survey items and were included in the final analytical sample
Arm/Group | Marshallese Adults in the U.S.
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 120
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 120

OUTCOME MEASURES:

1. Primary Outcome: Personal Preventative Behaviors to Decrease Risk of COVID-19 Exposure
Description: Participants will report behaviors they regularly engage in to lessen their risk of contracting COVID-19 (e.g., social distancing, wearing a mask, etc.). Participants were asked "Which of the following measures have you taken to prevent infection from COVID-19? (Select all that apply)"
Time Frame: Baseline
Population: N=117 due to missing data on this item for three participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Marshallese Adults in the U.S.
Number analyzed (Participants) | 117
Participants
  Hand washing for at least 20 seconds | 114
  Avoiding touching your eyes, nose, and mouth with unwashed hands | 112
  Use disinfectants to clean hands when soap and water not available for washing hands | 114
  Staying home when you are sick or when you have a cold | 109
  Asked family members or friends not to visit me: number analyzed (Participants) | 116
  Asked family members or friends not to visit me | 105
  Covering your mouth when you cough | 113
  Wearing a face mask | 115
  Physical distancing (keeping minimum 6 feet between you and others from outside your household) | 113
  Staying at home even if you do not feel sick | 99
  Disinfecting surfaces | 114

2. Primary Outcome: Workplace Preventative Actions to Decrease Risk of COVID-19 Exposure
Description: Participants will report specific steps taken by their employers to reduce risk of contracting COVID-19 (e.g., requiring remote work, mask mandates, etc.). Participants were asked to "Please check all of the following your workplace has done since the COVID-19 outbreak (Select all that apply)".
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Marshallese Adults in the U.S.
Number analyzed (Participants) | 120
Participants
  Required employees to work remotely or from home | 27
  Suggested employees work remotely or from home | 23
  Required employees to wear face masks | 73
  Suggested employees wear face masks | 41
  Provided employees with face masks | 58
  Required social distancing at work | 59
  Installed barriers / shields to reduce contact between employees and others | 31
  Taken employee temperatures before entering workplace | 61
  Asked COVID-19 screening questions of employees before entering workplace | 41
  Was tested for COVID-19 | 47
  None of these | 5
  Don't know/Not sure | 3

3. Secondary Outcome: Effects of COVID-19 on General Health Status
Description: Participants will be asked to rate their general health status compared with before the COVID-19 outbreak. Participants were asked "Compared to the time before the COVID-19 outbreak, is your physical health status better, worse, or about the same?"
Time Frame: Baseline
Population: N=119 due to missing data on this item for one participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Marshallese Adults in the U.S.
Number analyzed (Participants) | 119
Participants
  Better | 20
  About the same | 74
  Worse | 19
  Don't know/Not sure | 6

4. Secondary Outcome: Effects of COVID-19 on Access to Healthcare Services
Description: Participants will be asked to report ways in which the COVID-19 pandemic has disrupted access to healthcare (e.g., seeking routine care, getting necessary medications, etc.). Participants were asked "In what ways has the COVID-19 outbreak affected your overall healthcare? (Select all that apply)".
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Marshallese Adults in the U.S.
Number analyzed (Participants) | 120
Participants
  I did not go to healthcare appointments because of concern about entering my provider's office | 20
  My healthcare provider canceled appointment | 14
  My healthcare provider changed to phone or online visits | 20
  My healthcare provider told me to self-isolate or quarantine | 21
  None of these apply | 53
  Don't know/Not sure | 5

5. Secondary Outcome: Effects of COVID-19 on Dietary Habits
Description: Participants will be asked to compare their current dietary behaviors with before the COVID-19 outbreak. Participants were asked "How do you think your eating habits have changed compared to before the COVID-19 outbreak?"
Time Frame: Baseline
Population: N=119 due to missing data on this item for one participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Marshallese Adults in the U.S.
Number analyzed (Participants) | 119
Participants
  I feel that I am eating more healthy now than before the COVID-19 outbreak | 25
  I am eating about the same as before the COVID-19 outbreak | 41
  I feel that I am eating less healthy now than before the COVID-19 outbreak | 30
  I have not noticed | 18
  Don't know/Not sure | 5

6. Secondary Outcome: Effects of COVID-19 on Physical Activity Behaviors (Not Specifically for Exercise)
Description: After reporting how many times per week they engaged "in at least 30 minutes of physical activity that was not specifically for exercise (total minutes of continuous activity, including walking, yard work, construction work, etc.)", participants were then asked "Is this more, less or about the same as the number of days you participated in at least 30 minutes of physical activity that was not specifically for exercise (total minutes of continuous activity, including walking, yard work, construction work, etc.) in a typical week before the COVID-19 outbreak?"
Time Frame: Baseline
Population: N=119 due to missing data on this item for one participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Marshallese Adults in the U.S.
Number analyzed (Participants) | 119
Participants
  More | 27
  About the same | 52
  Less | 35
  Don't know/Not sure | 5

7. Secondary Outcome: Effects of COVID-19 on Physical Activity Behaviors (Specifically for Exercise)
Description: After reporting how many times per week they engaged "in at least 30 minutes of a specific exercise session (such as swimming, walking specifically for exercise, biking, etc.)", participants were then asked "Is this more, less or about the same as the number of days you participated in at least 30 minutes of a specific exercise session (such as swimming, walking specifically for exercise, biking etc.) in a typical week before the COVID-19 outbreak?"
Time Frame: Baseline
Population: N=119 due to missing data on this item for one participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Marshallese Adults in the U.S.
Number analyzed (Participants) | 119
Participants
  More | 17
  About the same | 56
  Less | 37
  Don't know/Not sure | 9

8. Secondary Outcome: Effects of COVID-19 on Weight
Description: Participants were asked to report changes in weight. Participants were asked "Have you noticed your weight change since the COVID-19 outbreak?"
Time Frame: Baseline
Population: N=119 due to missing data on this item for one participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Marshallese Adults in the U.S.
Number analyzed (Participants) | 119
Participants
  I have lost weight | 30
  I think I weigh about the same | 26
  I have gained weight | 34
  I have not noticed | 26
  Don't know/Not sure | 3

9. Secondary Outcome: Effects of COVID-19 on HbA1c (Glycated Hemoglobin)
Description: After reporting their most recent HbA1c reading, participants were then asked "How different was this HbA1c reading from your average HbA1c reading before the COVID-19 outbreak?"
Time Frame: Baseline
Population: Using survey skip logic, only those participants who selected "yes" to being previously diagnosed with type 2 diabetes were asked this question (n=13).
Measure: Count of Participants; unit: Participants
Arm/Group | Marshallese Adults in the U.S.
Number analyzed (Participants) | 13
Participants
  Higher | 2
  About the same | 5
  Lower | 3
  Don't know/Not sure | 3

10. Secondary Outcome: Barriers to Type 2 Diabetes Management Due to COVID-19
Description: Participants with type 2 diabetes were asked to report how the COVID-19 outbreak affected their access to type 2 diabetes supplies (insulin, needles, etc.). Participants were asked "Has the COVID-19 outbreak affected your level of access to the following? (Select all that apply)"
Time Frame: Baseline
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Marshallese Adults in the U.S.
Number analyzed (Participants) | 13
Participants
  Insulin | 2
  Needles | 1
  Blood glucose meters | 1
  Testing strips | 3
  Other diabetes medication | 0
  No issues to report | 9

11. Secondary Outcome: COVID-19 Screening
Description: Participants were asked to report whether they have been screened for COVID-19 and by what method (by phone, online, at work, etc.). Participants were asked "Were you screened for COVID-19? (Select all that apply)".
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Marshallese Adults in the U.S.
Number analyzed (Participants) | 120
Participants
  Yes, by phone | 9
  Yes, online | 7
  Yes, at a drive-through screening | 45
  Yes, at a healthcare clinic or hospital | 32
  Yes, at work | 27
  No | 28
  Don't know/Not sure | 6

12. Secondary Outcome: COVID-19 Testing
Description: Participants were asked to report whether they have been tested for COVID-19 and the results of the test. Participants were asked "Have you had the nose swab test for the virus that causes COVID-19? (Mark all that apply)"
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Marshallese Adults in the U.S.
Number analyzed (Participants) | 120
Participants
  No, I never tried to get tested | 20
  No, I tried to get tested but was not able to | 1
  Yes, and I am waiting for the results | 6
  Yes, and I tested negative | 54
  Yes, and I tested positive | 33
  Don't know/Not sure | 9

13. Secondary Outcome: COVID-19 Vaccine Willingness/Hesitancy
Description: Participants were asked to report whether they would accept a COVID-19 vaccine. Participants were asked "If a vaccine for COVID-19 were available today, what is the likelihood that you would get vaccinated?"
Time Frame: Baseline
Population: N=113 due to missing data on this item for seven participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Marshallese Adults in the U.S.
Number analyzed (Participants) | 113
Participants
  Extremely likely | 39
  Somewhat likely | 25
  Unlikely | 8
  Very unlikely | 9
  Don't know/Not sure | 32

14. Secondary Outcome: Trusted Sources of COVID-19 Information
Description: Participants were asked to report which sources of information they trust the most to stay informed about COVID-19. Participants were asked "What resource do you trust most for reliable information about COVID-19?"
Time Frame: Baseline
Population: N=117 due to missing data on this item for three participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Marshallese Adults in the U.S.
Number analyzed (Participants) | 117
Participants
  University of Arkansas for Medical Sciences | 12
  Community Clinic | 15
  Another healthcare organization | 1
  Dr. Sheldon Riklon's radio show or Facebook Live videos | 14
  News outlets | 4
  US Dept of Health (CDC, NIH, and other federal health agencies) | 40
  Your state Dept of Health | 17
  Marshallese Consulate/RMI Ministry of Health | 7
  Your pastor | 1
  Other | 1
  None | 1
  Don't know/Not sure | 4

15. Secondary Outcome: Effects of COVID-19 on Housing
Description: Participants were asked how COVID-19 has impacted their housing situation. Participants were asked "Please check all of the following that have happened to you since the COVID-19 outbreak".
Time Frame: Baseline
Population: N=118 due to missing data on this item for two participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Marshallese Adults in the U.S.
Number analyzed (Participants) | 118
Participants
  I have moved into a friend or family member's household | 3
  A friend or family member(s) have moved into my household | 12
  I became homeless (e.g., lived in a shelter, outside, or in a car) | 4
  None of these | 98
  Don't know/Not sure | 1

16. Secondary Outcome: Effects of COVID-19 on Employment
Description: Participants were asked how COVID-19 has impacted their employment. Participants were asked "In what ways has the COVID-19 outbreak affected your work? (Select all that apply)".
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Marshallese Adults in the U.S.
Number analyzed (Participants) | 120
Participants
  I lost my job permanently | 12
  I lost my job temporarily | 13
  I got a new job | 9
  I reduced my work hours | 27
  I increased my work hours | 4
  My job put me at increased risk of getting COVID-19 | 23
  I laid off employees | 4
  None of these apply | 27
  Don't know/Not sure | 5

17. Secondary Outcome: Effects of COVID-19 on Income
Description: Participants were asked how COVID-19 has impacted their income. Participants were asked "As a result of COVID-19, has your family income changed?"
Time Frame: Baseline
Population: N=119 due to missing data on this item for one participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Marshallese Adults in the U.S.
Number analyzed (Participants) | 119
Participants
  Yes, it increased our income | 3
  Yes, it decreased our income | 66
  No | 43
  Don't know/Not sure | 7

18. Secondary Outcome: Sources of Stress During COVID-19
Description: Participants were asked to report their greatest sources of stress from the COVID-19 outbreak (e.g., health concerns, financial concerns, etc.). Participants were asked "What have been your greatest sources of stress from the COVID-19 outbreak? (Select all that apply)"
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Marshallese Adults in the U.S.
Number analyzed (Participants) | 120
Participants
  Health concerns | 75
  Financial concerns | 90
  Impact on work | 75
  Impact on your child | 79
  Impact on your community | 61
  Impact on family members | 75
  Access to food | 59
  Access to baby supplies (e.g., formula, diapers, wipes) | 24
  Access to personal care products or household supplies | 43
  Access to medical care, including mental health care | 32
  Access to medical supplies (e.g., prescriptions, testing supplies, etc.) | 27
  Social distancing or being quarantined | 47
  Other | 5
  I am not stressed about the COVID-19 outbreak | 1
  Don't know/Not sure | 2

ADVERSE EVENTS:
Time Frame: Day of survey
Description: This was a one-time cross-sectional survey, so there was no contact with participants prior to, or after the completion of, the survey.
Arm/Group | Marshallese Adults in the U.S.
All-Cause Mortality (participants affected / at risk) | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT04474496/Prot_SAP_000.pdf